CLINICAL TRIAL: NCT01869543
Title: Benefits of High Efficiency Filtration to Children With Asthma
Brief Title: Asthma and Indoor-air: Reducing Exposures
Acronym: AIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 346123; 11-324 (Other Grant/Funding Number: California Air Resources Board)
Record Dates: First submitted 2013-04-03; First posted 2013-06-05 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stand Alone Air Cleaner-True/Sham (Experimental): The participant will have stand alone air cleaners placed in their home. They will have true filtration followed by sham filtration.
  Interventions: Other: Stand Alone Air Cleaner
- Stand Alone Air Cleaner-Sham/True (Experimental): Participants will have stand alone air cleaners placed in their homes. They will begin with sham filtration.
  Interventions: Other: Stand Alone Air Cleaner
- HVAC modification-True/Sham (Experimental): Participants will have their HVAC system modified to include high efficiency filtration. They will begin true filtration followed by sham filtration.
  Interventions: Other: HVAC Modification
- HVAC Modification-Sham/True (Experimental): Participants will have their HVAC system modified to include high efficiency filtration. They will begin sham filtration.
  Interventions: Other: HVAC Modification

INTERVENTIONS:
Other: Stand Alone Air Cleaner — This is an environmental intervention using a stand alone air cleaner designed to reduce the air pollution levels in the home.
  Arms: Stand Alone Air Cleaner-Sham/True; Stand Alone Air Cleaner-True/Sham
Other: HVAC Modification — This is an environmental intervention that modifies the home HVAC system to include high efficiency air filtration designed to reduce the air pollution levels in the home.
  Arms: HVAC Modification-Sham/True; HVAC modification-True/Sham

SUMMARY:
Two hundred moderate to severely asthmatic children (6-12 years) will be enrolled in a study to look at the effectiveness of high efficiency filtration of indoor air in homes on reducing asthma symptoms. One intervention group will have high efficiency filters or filtration systems installed in their central heating and air conditioning (HVAC) system. The second intervention group will have high efficiency portable air cleaners placed in the child's bedroom and in the main living area. Each participant will receive true air filtration for a year and a placebo for a year. During the placebo period a sham filter will be used that removes very little of the particles. Measures of health effects will include days of symptoms, unplanned utilization of the healthcare system for asthma-related illness, short-term medication use, peak exhaled flow, spirometry, and exhaled nitric oxide (eNO).

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years of age
* Living in Fresno, San Bernardino or Riverside Counties.
* Physician diagnosed asthma, as stated by the participant's caregiver.
* In the last six months, the child must have had asthma symptoms at least twice a week for several weeks in a row.

Exclusion Criteria:

* Children living in homes where more than 2 cigarettes are smoked per week in the home.
* Children that spend 2 or more nights per week in another home.
* Children living in homes that are planning on moving in the next 2 years.
* Children living in homes that keep their windows open most of the time.
* Children living in homes that have existing high efficiency filtration.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Days with asthma symptoms | Measured at 3, 6, 9, 12, 15, 18, 21, and 24 months
  The maximum number of days with symptoms, from a two-week recall period, will be determined every three months. The maximum number of days with symptoms will be defined as the largest value among the following three variables: (i) number of days with wheezing, tightness in the chest, or cough because of asthma, (ii) number of days that the child had to slow down or stop his/her play or activities because of asthma, wheezing or tightness in the chest, or cough, or (iii) number of nights that the child woke up because of asthma, wheezing or tightness in the chest, or cough.
  The seasonally adjusted mean difference in the number of symptom days between the true and sham filtration periods will be estimated using generalized linear mixed-effects regression models.

SECONDARY OUTCOMES:
Forced expiratory volume at one second, percent predicted (FEV1 % predicted) | Measured at 12 months and 24 months
  Lung function will be assessed using FEV1 % predicted. The adjusted mean difference in the FEV1% predicted between the true and sham filtration periods will be estimated using generalized linear mixed-effects regression models.
Forced vital capacity, percent predicted (FVC % predicted) | Measured at 12 months and 24 months
  Lung function will be assessed using FVC % predicted. The adjusted mean difference in the FVC% predicted between the true and sham filtration periods will be estimated using generalized linear mixed-effects regression models.
Peak Expiratory Flow Rate (PEFR) | Measured at 3, 6, 9, 12, 15, 18, 21, and 24 months
  Lung function will be assessed using morning peak expiratory flow rate (PEFR), averaged for all days over one-week testing periods. The seasonally adjusted mean difference in the PERF measure between the true and sham filtration periods will be estimated using generalized linear mixed-effects regression models.
Exhaled NO | Measure at 6, 12, 18, and 24 months
  The seasonally adjusted mean difference in the Exhaled NO between the true and sham filtration periods will be estimated using generalized linear mixed-effects regression models.
Days of missing school due to asthma | Measured at 3, 6, 9, 12, 15, 18, 21, and 24 months
  Days of missing school due to asthma will be expressed as a proportion of days of missing school versus the total number of school days during a two-week period. The seasonally adjusted mean difference in the proportion of missed school days between the true and sham filtration periods will be estimated using generalized linear mixed-effects regression models.
Days of missing work for parents due to child's asthma | Measured at 3, 6, 9, 12, 15, 18, 21, and 24 months
  Days of missing work due to child's asthma will be expressed as a proportion of days of missing work versus the total number of work days during a two-week period. The seasonally adjusted mean difference in the proportion of missed work days between the true and sham filtration periods will be estimated using generalized linear mixed-effects regression models.
Hospitalizations | Count during 1-year true filtration period and count during 1-year sham filtration period
  The number of overnight hospitalizations due to asthma will be assessed every 3 months during real and sham periods. Participants will report number of overnight hospitalizations due to asthma that occurred in the previous three months. The adjusted mean hospitalization incidence ratio between the true and sham filtration periods will be compared using mixed-effects Poison regression models.
Emergency Room Visits | Count during 1-year true filtration period and count during 1-year sham filtration period
  The number of emergency room visits due to asthma will be assessed every 3 months during real and sham periods. Participants will report number of emergency room visits due to asthma that occurred in the previous three months. The adjusted mean emergency room visit incidence ratio between the true and sham filtration periods will be compared using generalized mixed-effects regression models.
Unplanned Clinic Visits | Count during 1-year true filtration period and count during 1-year sham filtration period
  The number of unplanned clinic visits due to asthma will be assessed every 3 months during real and sham periods. Participants will report number of unplanned clinic visits due to asthma that occurred in the previous three months. The adjusted mean unplanned clinic visit incidence ratio between the true and sham filtration periods will be compared using generalized mixed-effects regression models.
Unplanned Steroid treatments | Count during 1-year true filtration period and count during 1-year sham filtration period
  The number of unplanned steroid treatments due to asthma will be assessed every 3 months during real and sham periods. Participants will report number of unplanned steroid treatments due to asthma that occurred in the previous three months. The adjusted mean unplanned steroid treatment incidence ratio between the true and sham filtration periods will be compared using generalized mixed-effects regression models.
Mini Pediatric Asthma Quality of Life Questionnaire (MiniPAQLQ) | Measured at 3, 6, 9, 12, 15, 18, 21, and 24 months
  The MiniPAQLQ has three composite domains, symptoms, emotional function, and activity limitation, each of which will be analyzed separately. The seasonally adjusted mean difference in each domain score between the true and sham filtration periods will be estimated using generalized linear mixed-effects regression models.
Allergy symptoms | Measured at 3, 6, 9, 12, 15, 18, 21, and 24 months
  Allergy symptoms during two week recall periods will be summarized into a composite score. The seasonally adjusted mean difference in the scores between the true and sham filtration periods will be using generalized linear mixed-effects regression models.
Respiratory disease | Count of incidents of respiratory disease during 1-year true filtration period and count during 1-year sham filtration period
  The number of incidents of respiratory disease will be assessed every 3 months during real and sham periods. Participants will report number of incidents of respiratory disease that occurred in the previous three months. The adjusted mean respiratory disease incidence ratio between the true and sham filtration periods will be compared using generalized mixed-effects regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Bennett, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis- Department of Public Health Sciences, Davis, California, United States